CLINICAL TRIAL: NCT01713751
Title: Surgical Site Infection Rates of Two Different Skin Closure Methods Used in Obese Patients After Cesarean Delivery
Brief Title: Surgical Site Infection Rates in Obese Patients After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASUOGRCT03-2012
Record Dates: First submitted 2012-10-14; First posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Cesarean section
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interrupted suturing Group (Active Comparator): Includes women who have their skin closed with interrupted mattress stitches using non-absorbable polypropylene [Prolene®]
  Interventions: Other: Interrupted suturing
- Subcuticular suturing Group (Active Comparator): Includes women who have their skin closed with subcuticular stitches using non-absorbable polypropylene [Prolene®].
  Interventions: Other: Subcuticular suturing

INTERVENTIONS:
Other: Interrupted suturing — Skin is closed with interrupted mattress stitches using non-absorbable polypropylene [Prolene®]
  Arms: Interrupted suturing Group
Other: Subcuticular suturing — Skin is closed with subcuticular stitches using non-absorbable polypropylene [Prolene®]
  Arms: Subcuticular suturing Group

SUMMARY:
The aim of this study is to determine the surgical site infection rate and patient satisfaction for subcuticular versus interrupted mattress suture in closure of skin at Cesarean delivery in obese patients.

DETAILED DESCRIPTION:
This is a randomized controlled trial conducted in Ain-Shams University Maternity Hospital on the period from March 2012 till August 2012. It included 130 pregnant women who underwent elective Cesarean section.

The aim of this study is to determine the surgical site infection rate and patient satisfaction for subcuticular versus interrupted mattress suture in closure of skin at Cesarean delivery in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: any female in childbearing period.
* Women planned for elective Cesarean section.
* Obese women (BMI ≥ 30 Kg/m2). Our study calculated the BMI of patients from their weight and height at admission, because the pre-pregnancy BMI was not available for all patients, and we hypothesized that the BMI at admission was a better indicator of body mass during the at-risk time for development of SSI than was the pre-pregnancy BMI.

Exclusion Criteria:

* Women who had concurrent overt infection (e.g.chorioamnionitis, pyelonephritis or chest infection).
* Women who had intraoperative events that may themselves predispose to perioperative infection (e.g. bowel injury, operative time more than 90 minutes, major blood loss).
* Women who had hemoglobin less than 10g/dl, preeclampsia, diabetes, rupture of membranes more than 12 hours, corticosteroid therapy.
* Patients who had non Pfannenstiel incision.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days after the operative procedure
  We used the definition devised and adopted by the Center for Disease Control and Prevention.

SECONDARY OUTCOMES:
Skin closure time | 15 minutes
Postoperative pain | 48 hours
  Measured by 10-cm visual analogue scale, zero being no pain and ten the worst possible pain
Short-term cosmetic wound outcome | 30 days
  We used Stony Brook Scar Evaluation Scale
Overall women satisfaction | 30 days
  A questionnaire is used to check the patient satisfaction (satisfied versus unsatisfied) regarding the wound appearance and wound related pain

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa I. Ibrahim, MD, Study Director — Assistant Professor of Obstetrics & Gynecology Faculty of Medicine, Ain Shams University

REFERENCES:
- [Derived] Ibrahim MI, Moustafa GF, Al-Hamid AS, Hussein MR. Superficial incisional surgical site infection rate after cesarean section in obese women: a randomized controlled trial of subcuticular versus interrupted skin suturing. Arch Gynecol Obstet. 2014 May;289(5):981-6. doi: 10.1007/s00404-013-3098-z. Epub 2013 Nov 24. PMID 24272023